CLINICAL TRIAL: NCT05952986
Title: A Randomized, Placebo-Controlled, Double-Blind, Phase I Study to Evaluate the Safety and Bridging Pharmacokinetics Profile of FB825 for Single Subcutaneous Administration in Healthy Adults
Brief Title: A Study to Evaluate the Safety and Bridging PK Profile of FB825 for Single Subcutaneous Administration in Healthy Adults
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Oneness Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FB825CLPK01
Record Dates: First submitted 2023-07-03; First posted 2023-07-19 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2023-07

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Injections, Subcutaneous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- cohort 1 (Experimental): FB825 300 mg or placebo with single SC administration in 3:1 ratio
  Interventions: Drug: FB825 or Placebo in subcutaneous route
- cohort 2 (Experimental): FB825 450 mg or placebo with single SC administration in 3:1 ratio
  Interventions: Drug: FB825 or Placebo in subcutaneous route
- cohort 3 (Experimental): 300 mg single IV administration
  Interventions: Drug: FB825 in intravenous route

INTERVENTIONS:
Drug: FB825 or Placebo in subcutaneous route — FB825 or placebo solution for SC injection
  Arms: cohort 1; cohort 2
Drug: FB825 in intravenous route — FB825 solution for IV infusion
  Arms: cohort 3

SUMMARY:
This is a randomized, placebo-controlled, and double-blind study to evaluate the safety and bridging PK profile of FB825 for single SC administration in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, nonsmoker (no use of tobacco or nicotine products within 3 months prior to screening), ≥18 and ≤55 years of age, with body mass index (BMI) ≥18.5 and ≤30.0 kg/m2 and body weight ≥50.0 kg.
* Healthy as defined by:

  1. the absence of clinically significant illness and surgery within 4 weeks prior to dosing.
  2. the absence of clinically significant history of neurological, endocrine, cardiovascular, respiratory, hematological, immunological, psychiatric, gastrointestinal, renal, hepatic, and metabolic disease.
  3. the Investigator judgment, based on clinical laboratory test results performed at screening.
* Female subjects of non-childbearing potential must be:

  1. post-menopausal (spontaneous amenorrhea for at least 12 months prior to dosing) with follicle-stimulating hormone (FSH) levels per laboratory standard; or
  2. surgically sterile at least 3 months prior to dosing.
* Sexually active female subjects of childbearing potential and non-sterile male subjects must be willing to use an acceptable contraceptive method for 167 days after dosing.
* Female subjects of childbearing potential who are sexually active with a non-sterile male partner (sterile male partners are defined as men vasectomized for at least 3 months prior to dosing) must be willing to use one of the following acceptable contraceptive methods for 167 days after dosing:

  1. simultaneous use of hormonal contraceptive or non-hormonal intrauterine device used for at least 4 weeks prior to dosing (must agree to use the same contraceptive for 167 days after dosing) and condom for the male partner;
  2. simultaneous use of diaphragm or cervical cap with spermicide and condom for the male partner, started at least 21 days prior to dosing;
  3. or total abstinence from heterosexual intercourse.
* Male subjects who are not vasectomized for at least 3 months prior to dosing and who are sexually active with a female partner of childbearing potential must be willing to use one of the following acceptable contraceptive methods for 167 days after dosing:

  1. simultaneous use of condom and hormonal contraceptive or non-hormonal intrauterine device used for at least 4 weeks prior to sexual intercourse for the female partner;
  2. simultaneous use of condom and a diaphragm or cervical cap with spermicide for the female partner;
  3. or total abstinence from heterosexual intercourse.
* Male subjects (including men who have had a vasectomy) with a pregnant partner must agree to use a condom for 167 days after dosing.
* Male subjects must be willing not to donate sperm for 167 days after dosing.
* Able to understand the study procedures and provide signed informed consent form (ICF) to participate in the study.

Exclusion Criteria:

* Any clinically significant abnormal finding at physical examination at screening.
* Clinically significant abnormal laboratory test results or positive serology test results for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, or human immunodeficiency virus (HIV) types 1 and 2 antibodies at screening.
* The subject has one or more of the following laboratory abnormalities at screening:

  1. Hemoglobin ≤10.5 g/dL
  2. Platelet count ≤99999 /mm3
  3. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) 2 × upper limit of normal [ULN] or higher
  4. Lipase 1.5 × ULN or higher
  5. Serum creatinine 1.5 × ULN or higher
  6. Any other clinically significant laboratory abnormality as judged by the Investigator
* Positive pregnancy test or lactating female subject.
* Positive urine drug screen, urine cotinine test, or alcohol breath test on Day -1.
* Known allergic reactions to FB825 or other related drugs, or to any excipient in the formulation.
* Clinically significant ECG abnormalities or vital signs abnormalities at screening.
* History of risk factors for torsade de pointes syndrome.
* History of drug abuse within 1 year prior to screening or recreational use of soft drugs within 1 month or hard drugs within 3 months prior to screening.
* History of alcohol abuse within 1 year prior to screening or regular use of alcohol within 6 months prior to screening that exceeds 7 units for women or 14 units for men of alcohol per week (1 unit = 340 mL of beer 5%, 140 mL of wine 12%, or 45 mL of distilled alcohol 40%).
* The subject lives in, has recently (within 6 months of screening) lived in or traveled to, or is planning to travel to, an area where parasitic infections are endemic. In cases of uncertainty, it can be judged by the Investigator prior to enrolling the subject in the study.
* The subject has clinically relevant, currently active or underlying gastrointestinal, cardiovascular, nervous system, psychiatric, metabolic, renal, hepatic, respiratory, inflammatory, immunological, endocrine, or infectious disease. This includes subjects with asthma, eosinophilic disease of any origin, IgE abnormalities, or urticaria of all types.
* The subject has a clinically significant history, as determined by the Investigator, of drug allergies or hypersensitivity such as, but not limited to, sulfonamides and penicillins, or a drug allergy witnessed in a previous study with experimental drugs.
* The subject has any history of a previous anaphylactic reaction.
* The subject has used a concomitant medication, including over-the-counter (OTC) products, herbal medications, dietary supplements, and vitamin supplements within 14 days before Day -1.
* The subject has received any immunoglobulin products or blood products within 6 months of Day -1 or has any previous participation in a clinical research study involving the administration of FB825.
* Participation in a clinical research study involving the administration of an investigational or marketed drug or device within 30 days (or 5 half-lives, whichever is longer) prior to Day -1, administration of a biological product in the context of a clinical research study within 90 days prior to Day -1, or concomitant participation in an investigational study involving no drug or device administration.
* Donation of plasma within 2 months prior to dosing or donation or loss of 500 mL or more of whole blood within 2 months prior to dosing.
* Subject has the presence of tattoos, sunburn, or other skin disturbances on injection/infusion site which may interfere with a medical assessment of the injection/infusion site both prior to and following dosing.
* The subject is a member of the site study team.
* The subject has any condition that, in the opinion of the Investigator, would compromise the study or the well-being of the subject or prevent the subject from meeting or performing study requirements.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2023-05-03 (Actual); Primary Completion 2024-03-26 (Estimated); Study Completion 2024-03-26 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse event | 24 months
  Safety will be reported based on Protocol defined AEs.
  For the purpose of this protocol, an AE will be defined as any untoward medical occurrence in a subject during the study.
AUC0-inf | 19 months
  Area under the concentration-time curve from time zero to infinity, (extrapolated) will be assessed
AUC0-t | 19 months
  Area under the concentration-time curve from time zero until the last observed concentration will be assessed
Cmax | 19 months
  Maximal observed concentration will be assessed

SECONDARY OUTCOMES:
absolute bioavailability factor | 19 months
  Absolute bioavailability factor will be assessed
Tmax | 19 months
  Time of observed Cmax will be assessed
T½ el | 19 months
  Elimination half-life will be assessed
Kel | 19 months
  Elimination rate constant will be assessed
CL/F | 19 months
  Apparent clearance (for SC administration) will be assessed
Vd/F | 19 months
  Apparent volume of distribution (for SC administration) will be assessed
CL | 19 months
  Total body clearance (for IV infusion) will be assessed
Vd | 19 months
  Volume of distribution (for IV infusion) will be assessed
Residual area | 19 months
  Calculated as 100*(1- (AUC0-last / AUC0-inf))
The effect of FB825 in immunogenicity | 19 months
  Immunogenicity will be reported based on anti-drug antibody concentration.

CONTACTS AND LOCATIONS:
Locations (1):
- Phase I center, Anaheim, California, United States